CLINICAL TRIAL: NCT07326878
Title: A Single-center, Randomized, Double-blind, and Placebo Controlled Phase Ⅰ Clinical Trial of the Safety and Preliminary Immunogenicity of Enterovirus Type71 - Coxsackievirus Type A16 Bivalent Vaccine in People Aged 6 Months to 59 Years
Brief Title: Phase I Clinical Trial of Enterovirus Type71 - Coxsackievirus Type A16 Bivalent Vaccine
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: EV71-CA16-101
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Hand, Foot and Mouth Disease (HFMD); HFMD; Hand, Foot and Mouth Disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Intervention Model Description: The dose escalation principle within each age group is from low to high doses, the sequential enrollment principle between different age groups is from adults to children.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low-dose experimental group (Experimental): Participants aged 18~59 years old, 6~17years old, 6months old~5 years old
  Interventions: Biological: Low Dose Enterovirus Type71 - Coxsackievirus Type A16 bivalent vaccine, inactivated (human diploid cell)
- medium-dose experimental group (Experimental): Participants aged 18~59 years old, 6~17years old, 6months old~5 years old
  Interventions: Biological: Medium Dose Enterovirus Type71 - Coxsackievirus Type A16 bivalent vaccine, inactivated (human diploid cell)
- high-dose experimental group (Experimental): Participants aged 18~59 years old, 6~17years old, 6months old~5 years old
  Interventions: Biological: High Dose Enterovirus Type71 - Coxsackievirus Type A16 bivalent vaccine, inactivated (human diploid cell)
- Placebo control group (Placebo Comparator): Participants aged 18~59 years old, 6~17years old, 6months old~5 years old
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low Dose Enterovirus Type71 - Coxsackievirus Type A16 bivalent vaccine, inactivated (human diploid cell) — Low-dose vaccine，dosage and immunization procedure: 0.1 ml/dose, 2 doses, 28-day interval
  Arms: low-dose experimental group
Biological: Medium Dose Enterovirus Type71 - Coxsackievirus Type A16 bivalent vaccine, inactivated (human diploid cell) — Medium-dose vaccine，dosage and immunization procedure: 0.1 ml/dose, 2 doses, 28-day interval
  Arms: medium-dose experimental group
Biological: High Dose Enterovirus Type71 - Coxsackievirus Type A16 bivalent vaccine, inactivated (human diploid cell) — High-dose vaccine，dosage and immunization procedure: 0.1 ml/dose, 2 doses, 28-day interval
  Arms: high-dose experimental group
Biological: Placebo — Placebo，dosage and immunization procedure: 0.1 ml/dose, 2 doses, 28-day interval
  Arms: Placebo control group

SUMMARY:
This is a randomized, double-blinded, placebo-controlled phase I clinical trial to evaluate the safety and preliminary immunogenicity of the Enterovirus Type71 - Coxsackievirus Type A16 bivalent vaccine in subjects ( aged 6 months to 59 years ).

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blinded, placebo-controlled phase I clinical trial in which three dose levels of the Enterovirus Type71 -Coxsackievirus Type A16 bivalent vaccine will be evaluated the safety and preliminary immunogenicity in subjects aged 6 months to 59 years. A total of 144 participants will be enrolled, including 48 adults (aged 18-59 years), 48 adolescents (aged 6-17 years), and 48 children (aged 6 months-5 years). Participants will be randomized into vaccine group and placebo group in a 3:1 ratio, and receive two doses of vaccine or placebo according to the 0- and 28-day immunization schedule.The dose escalation principle within each age group is from low to high doses, and the sequential enrollment principle between different age groups is from adults to children.

Primary endpoints are the occurrence of safety events after vaccination including the incidence of adverse events within 30 minutes/7 days/28 days after each dose, as well as the incidence of serious adverse events within 12 months after the final dose which will be defined as the secondary safety endpoint. Besides, the secondary immunogenicity endpoints are the geometric mean titers, geometric mean fold increases, seropositive rates, and seroconversion rates of anti-EV71 neutralizing antibodies and anti-CA16 neutralizing antibodies 28 days after the final dose.

ELIGIBILITY:
Inclusion Criteria:

* Age Requirement: volunteers aged 6 months and 59 years.
* Provision of Legal Identification: volunteers and their legal guardians or appointed representatives must provide valid legal identification documents.
* Informed Consent: participants, legal guardians, or appointed representatives of volunteers must have the capacity to understand the informed consent document and the research process, voluntarily participate, sign the informed consent form, and be able to comply with the requirements in the study as well as complete relevant visits on time.
* 6~23months old: term delivery (gestational week 37 weeks ~ 42 weeks at birth), 2500g ≤ birth weight ≤ 4000g.
* Requirements for contraception: agree to take contraception actions in 12 months.
* Temperature Requirement: axillary body temperature is less than 37.3°C.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will be not eligible for enrollment.

* Subjects who have been allergic to any component of the vaccine in the past, or have any history of vaccine allergy or suspected allergy or other serious adverse reactions, such as urticaria, respiratory distress, and angioedema.
* History of taking administration of a non-SARS-CoV-2 inactivated vaccine or subunit vaccine within 7 days before enrollment, or any live attenuated vaccine or SARS-CoV-2 vaccine within 14 days before enrollment.
* Subjects with convulsion, epilepsy, encephalopathy, psychiatric history or family history.
* Known to have serious congenital malformations, developmental disorders, genetic defects or abnormal growth and development, or clinically diagnosed serious chronic diseases, including but not limited to neurological, cardiovascular, blood and lymphatic system, immune system, kidney, liver, gastrointestinal, respiratory system, metabolism and bone diseases and a history of malignant tumors.
* Subjects are acutely ill or in the acute phase of a chronic illness within 3 days before vaccination.
* Subjects with a hereditary bleeding tendency or coagulopathy, or a history of bleeding disorders.
* Subjects who intolerance to venipuncture and with a history of needle- or blood-induced syncope.
* History of surgical removal of the spleen or other vital organs for any reason.
* Donation or loss of blood (≥400 mL), receipt of blood products, or receipt of blood transfusion within the 3 months before enrollment.
* Use of any investigational or unregistered product (drug, vaccine, biological product, or device) other than a study vaccine within 3 months before enrollment or planned for use during the study.
* Have treatment with immunosuppressive agents within 6 months before enrollment, such as long-term systemic glucocorticoid therapy (e.g., prednisone or a similar drug for more than 2 consecutive weeks within 6 months), but topical use (e.g., ointments, eye drops, inhalers, or nasal sprays) was allowed. Topical use should not exceed the recommended dose on the label or have any signs of systemic exposure.
* History of any EV71 antigen-containing vaccination, whether commercially available or investigational.
* Subjects with history of hand, foot, and mouth disease.
* Subjects with abnormal vital signs with clinical significance.
* Subjects who do not meet the criteria for good health based on comprehensive physical examination, including: (1) abnormal vital signs with clinical significance; (2) clinical laboratory testing shows laboratory abnormalities and with clinical significance (applicable only to subjects aged 2 years and above).
* Have been diagnosed with an infectious disease that may interfere with the conduct or completion of the study, such as active tuberculosis, viral hepatitis, human immunodeficiency virus (HIV) infection, etc.
* Females with positive pregnancy test results.
* Females who are lactating, or subjects who plan to conceive or to donate sperm or ova from the time of signing the informed consent form until 12 months after completion of the full vaccination schedule (applicable only to subjects aged 18 to 59 years).
* Subjects with a history of abnormal birth delivery, birth asphyxia, neurological impairment, or clinically diagnosed pathological jaundice (applicable only to subjects aged 6 to 23 months).
* Subjects deemed by the investigator to be unsuitable for participation in the study.

Ages: 6 Months to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Safety index - incidence of adverse events | 0- 30 minutes/Day 0 to 7 days/Day 0 to 28 days after each dose
  Incidence of adverse events after each dose vaccination

SECONDARY OUTCOMES:
Safety index - incidence of serious adverse events | From the beginning of the vaccination up to12 months after the last vaccination completed
  Incidence of serious adverse events/adverse reactions after vaccination
Immunogenicity index-Seroconversion rates | Between baseline and Day 28 after full vaccination
  The seroconversion rates of anti-EV71 neutralizing antibodies and anti-CA16 neutralizing antibodies after the end of the entire vaccination course.
Immunogenicity index - Geometric mean titer (GMT) | Day 28 after full vaccination
  The GMT of anti-EV71 neutralizing antibodies and anti-CA16 neutralizing antibodies 28 days after the end of the entire vaccination course.
Immunogenicity index - Geometric mean fold increases (GMFI) | Between baseline and Day 28 after full vaccination
  The GMFI of anti-EV71 neutralizing antibodies and anti-CA16 neutralizing antibodies after the end of the entire vaccination course.
Immunogenicity index-Seropositive rates | Day 28 after full vaccination
  The seropositive rates of anti-EV71 neutralizing antibodies and anti-CA16 neutralizing antibodies 28 days after the end of the entire vaccination course.

CONTACTS AND LOCATIONS:
Overall Officials: Xian Yu, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No